CLINICAL TRIAL: NCT01684891
Title: Single-center, Open Label, Multiple Dose Study to Investigate the Pharmacokinetics of RG1662 Given BID Over 28 Days, and in Addition, the Excretion and Metabolism of [13C]-Labelled IV Microdoses and an Oral [14C]-Labelled Dose of RG1662 in Healthy Male Volunteers
Brief Title: A 28-Day Pharmacokinetics Study of RG1662 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: WP28214; 2012-001434-34 (EudraCT Number)
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

ARMS (1):
- RG1662 (Experimental)
  Interventions: Drug: RG1662

INTERVENTIONS:
Drug: RG1662 — multiple doses of RG1662

SUMMARY:
This is a single-center, open label, multiple dose study to investigate the pharmacokinetics of RG1662 given twice daily over 28 days, and in addition, the excretion and metabolism of [13C]-labeled IV microdoses and an oral [14C]-labeled dose of RG1662 in healthy male volunteers. The anticipated time of study treatment is 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* Volunteers who are surgically sterilized or who do not intend to father children in the future
* Absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, serology and urinalysis
* Body mass index (BMI) between 18 and 30 kg/m2 inclusive
* Volunteers and their partners of childbearing potential must use two medically approved methods of contraception (e.g. hormonal contraception, IUD, barrier contraception), one of which must be a barrier method, for the duration of the study and for 3 months after last drug administration

Exclusion Criteria:

* If capable of reproduction, unwilling to use an effective form of contraception
* Suspicion of regular consumption of drug of abuse
* Positive result on hepatitis B (HBV), hepatitis C (HCV), or HIV 1 and 2
* Clinically relevant ECG abnormalities at screening
* Family history of congenital long QT syndrome or known congenital arrhythmia
* Systolic blood pressure greater than 140 or less than 90 mm Hg, and diastolic blood pressure greater than 90 or less than 50 mm Hg. Resting Pulse Rate greater than 90 or less than 45 beats per minute
* Any other clinical relevant clinical abnormalities
* Participation in an investigational drug or device study within 90 days prior to screening
* Donation of more than 500 mL of blood within three months prior to screening
* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the volunteer in this study

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Area under the concentration time curve (AUC) | Selected Days between 1 and 28
Pharmacokinetics: maximum serum concentration | Selected Days between 1 and 28
Pharmacokinetics: Clearance of 13C-RG1662 | Days 1 and 28
Pharmacokinetics: Bioavailability of 13C-RG1662 | Days 1 and 28

SECONDARY OUTCOMES:
Amount of drug excreted in urine over the sampling interval | Days 1 to 15
Amount of drug excreted in the feces over the sampling interval | Pre-dose, days 1 to 15
Incidence of adverse events | Up to approximately 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Zuidlaren, Netherlands